CLINICAL TRIAL: NCT05585333
Title: Photobiomodulation Therapy for Facial Paralysis Over 8 Weeks: An Open-Label Pilot, Non-concurrent Control Study
Brief Title: Photobiomodulation Therapy Treatment on Facial Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBMT-FP-2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-02

CONDITIONS: Facial Paralysis
Keywords: Facial paralysis; photobiomodulation; ENoG; EMG; HB grading
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Group (Experimental): Treatments were performed with MLS laser (Mphi laser, ASA Srl, Italy). MLS laser is a class IV NIR laser with two synchronized sources (laser diodes). The first one is a pulsed laser diode, emitting at 905 nm, with 25 W peak power. The second laser diode (808 nm) was operated in a continuous mode with power 1 W. Both of the laser beams were synchronized, the locked waves work within the range 1-2000 Hz.
  Interventions: Device: MLS laser
- Control Group (No Intervention)

INTERVENTIONS:
Device: MLS laser — Treatments were performed with MLS laser (Mphi laser, ASA Srl, Italy). MLS laser is a class IV NIR laser with two synchronized sources (laser diodes). The first one is a pulsed laser diode, emitting at 905 nm, with 25 W peak power. The second laser diode (808 nm) was operated in a continuous mode with power 1 W. Both of the laser beams were synchronized, the locked waves work within the range 1-2000 Hz.
  Arms: Photobiomodulation Group

SUMMARY:
Objective: Facial paralysis can be caused by a variety of etiological factors, complete palsy continues for two months, the chance of full recovery is reduced to zero. The aim of this study was to evaluate the effectiveness of photobiomodulation therapy (PBMT) in the in patients undergoing facial paralysis over 8 weeks.

Methods: This study was an open-label, not concurrent control study including 54 patients that underwent facial paralysis over 8 weeks. Patients were assigned to the PBMT group and control group, with 27 patients in each group. Laser treatments were applied 3 days a week after recruited. PBMT was delivered using a class IV Multi-wave Locked System that combines with a simultaneous 808 nm continuous emission and 905 nm pulse emission and the maximum peak power was 25 W. Clinical outcome measure comprised the House-Brackmann grading system, Facial Clinimetric Evaluation Scale (FaCE), Sunnybrook facial grading scale (SBFG), and electrophysiological testing, including Electroneuronography (ENoG), Electromyography (EMG) and Blink Reflex. All the measurements were collected at the first day and at the end of study. All reported P values were two-sided and were declared statistically significant when less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

- (1) adults over 18 years of age and under 65 years of age. (2) had not received medicine, such as prednisolone. (3) had history of Bell's palsy, Ramsay Hunt syndrome, traumatic facial paralysis and history of otological surgery.

(4) Disease duration longer than two months.

Exclusion Criteria:

- (1) Complete facial paralysis (HB 6). (2) Greater than 90% denervation on ENoG. (3) No voluntary EMG activity. (4) No latency of early (R1) and late (R2, R2') components in blink reflex. (5) Serious mental illness or social problems, and neurological disorders. (6) Systemic disease, such as severe diabetes, malignant tumors and other serious consumptive diseases.

(7) Planning for pregnancy, in pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
The House-Brackmann Facial Nerve Grading System | Change from Baseline number of pathological HB grading at 6-months in post-therapy.
  The House-Brackmann facial nerve grading system (HB grading) is based on a 6-grade score that offers a gross evaluation of facial motor function and includes the evaluation of sequelae. The prognoses of patients with House-Brackmann grade I or grade II were considered good, and the prognoses of those with grade 3 or higher were considered poor.
The Sunnybrook Facial Grading System | Change from Baseline scores of SB grading at at 6-months in post-therapy.
  The Sunnybrook facial grading system (SB grading) is 13-items, self-reported questionnaire that used to evaluate the facial movement of patients. Among the overall 13 items of question, 3 items are resting symmetry, 5 items are symmetry of voluntary movement, and 5 items are synkinesis. Lower scores of Sunnybrook equate to greater severity of facial paralysis symptoms.
Facial Clinimetric Evaluation Scale | Change from Baseline scores of FaCE at at 6-months in post-therapy.
  The Facial Clinimetric Evaluation Scale (FaCE) is 15-items, self-reported questionnaire that used to assess facial impairment and disability after facial paralysis. Among the overall 15 items of question, FaCE grouped into six independent domains: social function, facial movement, facial comfort, oral function, eye comfort, and lacrimal control. Each using a five-item Likert scale. A participant circles the most appropriate response to a given statement, whereby 1 corresponds to the lowest function and 5 corresponds to the highest function. The total score is ranged 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Electroneuronography (ENoG) | Change from Baseline amplitude and potential of CAMP and the numbers of pathological ENoG at at 6-months in post-therapy.
  The goal of the Electroneurography (ENoG) testing is to measure the amount of neural degradation that has occurred distal to the site of facial nerve injury by measuring the muscle response to an electrical stimulus. The testing of ENoG involves recording the compound muscle action potential (CAMP) of the mimetic muscles, including Orbicularis oculi, Frontalis muscle, Orbicularis oris and Zygomaticus muscle.
  ENoG is performed first on the healthy side of the face and then on the affected side. Nerve damage or nerve fiber degeneration leads to a decrease or loss of the CAMP. The amplitude of the CAMP on the affected side is compared to the CAMP of the healthy side and expressed as percent (amplitude of the paralyzed side divided by the amplitude of the normal side). A side difference of 30% or bigger is considered pathologic.
Electromyography (EMG) | Change from Baseline amplitude and duration of MUAPs at at 6-months in post-therapy.
  EMG is an electrophysiologic measures that indirectly quantify facial nerve function by recording motor unit action potentials (MUAPs) in the muscle of Musculus depressor angulli oris, Frontalis muscle and Orbicularis oris. MUAPs are the spikes in electrical activity generated when a motor unit fires. A motor unit consists of a motor neuron and the corresponding muscle fibers innervated by the neuron.
Blink Reflex | Change from Baseline number of pathological Blink Reflex at 6-months in post-therapy.
  The blink reflex test is to measures the facial nerve since the blink reflex delivers information on facial nerve function with normal trigeminal function. Blink reflex testing involves electrical stimulation of the supraorbital nerve on the affected side combined with a 2-channel simultaneous sEMG recording from both orbicularis oculi muscles. The exit of the supraorbital nerve in the supraorbital foramen is palpated on the rim of the orbit. Stimulation with 10-20 mA and 0.2 ms duration is used to produce a constant reflex.
  In blink reflex testing, two responses, R1 and R2, are analyzed. R1 is the fast ipsilateral response of the orbicularis oculi muscle with a latency of about 10-12 ms. The second bilateral response R2 has a latency of about 30-41 ms.
  The R2 latency differences between both sides higher than 5-8 ms is considered pathologic.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Wu D, Zhao YL, Sun JY, Dai RJ, Cao K, Qu RK, Wang Y, Wu YQ. A Nonrandomized Trial of the Effects of Near-Infrared Photobiomodulation Therapy on Bell's Palsy with a Duration of Greater Than 8 Weeks. Photobiomodul Photomed Laser Surg. 2023 Sep;41(9):490-500. doi: 10.1089/photob.2023.0056. PMID 37738368